CLINICAL TRIAL: NCT07072156
Title: The Effect of Stress Ball Use on Stress, Anxiety, and Vital Signs in Patients Undergoing Chemotherapy for Breast Cancer
Acronym: Stressball
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Bedriye Cansu DEMİRKIRAN, assistant professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Stresballbreastca
Record Dates: First submitted 2025-07-07; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy; Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Stress Ball; breast cancer; stress; Anxiety; Vital Signs
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Stress Ball Group
  First Interview: Consent is obtained; group allocation is done.
  Pre-test: Patient information form, DT, STAI, and vital signs are assessed.
  Intervention: Stress ball use for 15-20 minutes during chemotherapy.
  Post-test: Same measurements are repeated.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress ball group (Experimental): Stress Ball Group
  First Interview: Consent is obtained; group allocation is done.
  Pre-test: Patient information form, DT, STAI, and vital signs are assessed.
  Intervention: Stress ball use for 15-20 minutes during chemotherapy.
  Post-test: Same measurements are repeated.
  Interventions: Other: Stress ball
- Control Group (No Intervention): Same steps as above, but no intervention; only routine treatment is provided.

INTERVENTIONS:
Other: Stress ball — First Interview: Consent is obtained; group allocation is done.
  Pre-test: Patient information form, DT, STAI, and vital signs are assessed.
  Intervention: Stress ball use for 15-20 minutes during chemotherapy.
  Post-test: Same measurements are repeated.
  Arms: Stress ball group

SUMMARY:
AIM This study aims to investigate the effects of stress ball use on stress, anxiety, and vital signs in patients receiving chemotherapy for breast cancer.

METHOD This study will be conducted with 50 breast cancer patients receiving chemotherapy at the Outpatient Chemotherapy Unit of Rize Training and Research Hospital, using a randomized controlled experimental design. Simple randomization will be used for group assignment. Data will be collected using a Breast Cancer Patient Information Form, Distress Thermometer, and State Anxiety Inventory. It is planned that data will be collected both before and after the chemotherapy session.

ORIGINALITY / SCIENTIFIC CONTRIBUTION To date, no study has been found in the literature evaluating the effects of stress balls on stress, anxiety, and vital signs in breast cancer patients undergoing chemotherapy. Therefore, this project is considered original and is expected to contribute to both national and international scientific literature. If successful, the project will provide evidence for a new non-pharmacological intervention that is easy to use during chemotherapy sessions and can help improve patients' stress, anxiety, and vital signs. Patients may experience more comfort and better treatment compliance during chemotherapy.

EXPECTED OUTCOMES It is expected that the use of a stress ball will have a positive effect on reducing stress and anxiety levels and improving vital signs in breast cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
METHOD This study is planned as a single-blind, randomized controlled experimental design. It will be conducted with breast cancer patients receiving chemotherapy at Rize Training and Research Hospital's Chemotherapy Unit.

POPULATION AND SAMPLE The study population consists of breast cancer patients receiving chemotherapy at the aforementioned hospital during the research period. Since no previous study has evaluated the effect of stress ball use on stress, anxiety, and vital signs in this population, the sample size was calculated using Cohen's large effect size (d = 0.80) via the G*Power 3.1.9.7 program. With α = 0.05 and power = 80%, the minimum required sample size was found to be 42. To account for possible data loss, 20% more participants will be included. Therefore, 25 patients will be assigned to each group, totaling 50 participants. The study will be reported in accordance with the CONSORT guidelines for randomized controlled trials.

INCLUSION CRITERIA Stage 2A-2B breast cancer

Receiving neoadjuvant chemotherapy

On a chemotherapy protocol administered every 21 days

Receiving second or subsequent chemotherapy cycle

No migraine, vertigo, active nausea, vomiting, or headache

No history of seizures

No primary or metastatic brain cancer

No visual, hearing, or cognitive impairment

Age 18 or older

No communication barriers

Voluntary participation

EXCLUSION CRITERIA Cancer types other than breast cancer

Unilateral or bilateral mastectomy

Any condition preventing hand use (e.g., pain, fracture, open wound)

IV access in both arms

Psychiatric diagnosis

Diagnosed anxiety disorder or current anti-anxiety medication use

WITHDRAWAL CRITERIA Patient requests to withdraw

Change in institution or city

Any illness developed during the intervention

Patient's death

RANDOMIZATION Patients meeting inclusion criteria and consenting to participate will be randomized into two groups using simple randomization via Excel's RAND function. Patients assigned even numbers will be placed in the stress ball group, and those with odd numbers in the control group.

BLINDING To minimize bias, both the researcher and the statistician will be blinded. Randomization will be performed by a researcher not involved in data collection. While the researcher administering the intervention will be aware of group allocation, data entry into SPSS will label groups as "Group 1" and "Group 2" without revealing the group type to the statistician.

IMPLEMENTATION OF THE RESEARCH Fifty eligible and consenting patients will be selected. After collecting pre-test data (prior to chemotherapy), patients in the intervention group will receive a stress ball following premedication. They will be instructed to focus on and squeeze the ball for 15-20 minutes during chemotherapy. The control group will continue with routine treatment and care. Post-test data will be collected after the chemotherapy session.

STRESS BALL DETAILS The stress ball is made of high-quality silicone, regaining its shape after squeezing. The ball used in this study is medium firmness (blue), elliptical, and 6 cm in diameter, suitable for adult use. Patients will be taught how to use the stress ball, including coordinated breathing techniques (inhale when squeezing, exhale when releasing). Stress balls will be given to intervention group patients to keep. Control group patients may request a ball after the study concludes.

DATA COLLECTION TOOLS Data will be collected using the Breast Cancer Patient Information Form, Distress Thermometer, and State Anxiety Inventory. Pre- and post-chemotherapy session measurements are planned.

Breast Cancer Patient Information Form:

Includes 11 items regarding age, marital status, education, economic status, employment, smoking and alcohol use, disease duration and stage, presence of chronic illness, and family history of cancer.

Distress Thermometer (DT):

Assess psychosocial distress in cancer patients. It uses a scale from 0 (no distress) to 10 (extreme distress). Scores ≥4 are considered clinically significant. Turkish validity and reliability studies were conducted by Özalp et al.

State Anxiety Inventory (STAI):

This study uses the state anxiety subscale to assess anxiety triggered by specific situations. It consists of 20 items scored on a 4-point Likert scale, where total scores range from 20 to 80. Higher scores indicate greater anxiety.

DATA ANALYSIS Data will be analyzed using SPSS version 26. Descriptive statistics (number, percentage, mean, standard deviation) will be used. For within-group comparisons: paired samples t-test (normal distribution) or Wilcoxon test (non-normal). For between-group comparisons: independent samples t-test (normal) or Mann-Whitney U test (non-normal). A p-value of <0.05 will be considered statistically significant.

STUDY FLOWCHART SUMMARY Stress Ball Group

First Interview: Consent is obtained; group allocation is done.

Pre-test: Patient information form, DT, STAI, and vital signs are assessed.

Intervention: Stress ball use for 15-20 minutes during chemotherapy.

Post-test: Same measurements are repeated.

Control Group

Same steps as above, but no intervention; only routine treatment is provided.

LIMITATIONS This study is limited to 50 breast cancer patients receiving chemotherapy at the outpatient chemotherapy unit of Rize Training and Research Hospital.

BUDGET JUSTIFICATION 25 stress balls for the intervention group

5 spare stress balls

10 stress balls for the control group (to be given post-study upon request)

RESEARCH FACILITIES Access to 50 breast cancer patients at Rize Training and Research Hospital's Outpatient Chemotherapy Unit

Researcher computers provided by affiliated universities

Hospital devices (blood pressure monitor and pulse oximeter) for vital sign measurements

Stress balls to be purchased with project funds

ELIGIBILITY:
Inclusion Criteria:

* Stage 2A-2B breast cancer
* Receiving neoadjuvant chemotherapy
* On a chemotherapy protocol administered every 21 days
* Receiving second or subsequent chemotherapy cycle
* No migraine, vertigo, active nausea, vomiting, or headache
* No history of seizures
* No primary or metastatic brain cancer
* No visual, hearing, or cognitive impairment
* Age 18 or older
* No communication barriers
* Voluntary participation

Exclusion Criteria:

* Cancer types other than breast cancer
* Unilateral or bilateral mastectomy
* Any condition preventing hand use (e.g., pain, fracture, open wound)
* IV access in both arms
* Psychiatric diagnosis
* Diagnosed anxiety disorder or current anti-anxiety medication use

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Distress Thermometer (DT): | 1 per month for 3 months
  It assesses the state anxiety an individual feels due to the stressful situation they are in, their predisposition to this anxiety, and the trait anxiety that generally characterizes the situations they find themselves in as stressful. The total score on the scale ranges from 20 to 80, with higher scores indicating higher anxiety levels and lower scores indicating lower anxiety levels.

SECONDARY OUTCOMES:
State Anxiety Inventory (STAI): | 1 per month for 3 months
  It assesses the state anxiety an individual feels due to the stressful situation they are in, their predisposition to this anxiety, and the trait anxiety that generally characterizes the situations they find themselves in as stressful. The total score on the scale ranges from 20 to 80, with higher scores indicating higher anxiety levels and lower scores indicating lower anxiety levels.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol